CLINICAL TRIAL: NCT00477568
Title: Back Pain Prevalence in Wheelchair Users and Associated Risk Factors
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Collaborators: Mallorca Institute of Social Affairs (Other Government)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Other Study IDs: FK-R-14
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Back Pain
Keywords: Wheelchair users; Back pain; Prevalence; Risk factors
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to determine the prevalence of back pain in permanent wheelchair users (excludes transitory users) in different regions of Spain. Another study objective is the identification of risk factors for back pain in this population. Data collection will be by means of a structured questionnaire which will be validated in a previous pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Adults with established disability;
* Permanent wheelchair users;
* Having physical and intellectual ability to answer questionnaire.

Exclusion Criteria:

* Transitory wheelchair users;
* Diagnosis of inflammatory rheumatic disease, cancer, systemic infection;
* Red flags for systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wheelchair users who do so on a constant basis (not occasional).
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2007-11; Primary Completion 2015-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Unidad de la Espalda Kovacs, Hospital Universitario HLA-Moncloa; Juan Noguera, MD, Principal Investigator — Instituto de Asuntos Sociales y Deportes de Mallorca, Palma de Mallorca, Spain
Locations (2):
- Spain (2):
  - Fundación Kovacs, Palma de Mallorca, Balearic Islands
  - Instituto de Asuntos Sociales y Deportes de Mallorca, Palma de Mallorca, Balearic Island